CLINICAL TRIAL: NCT06655688
Title: The Effect of Acceptance and Commitment Therapy on Self-Stigmatization, Coping With Stress and Psychological Resilience Levels of Family Members After First Psychotic Attack Diagnosis
Brief Title: Acceptance and Commitment Therapy (ACT) for Family Members After a First Psychotic Attack
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Duygu Özer, PhD, Asst. Prof., Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BARU-SBF-DO-1
Record Dates: First submitted 2024-10-19; First posted 2024-10-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-10

CONDITIONS: First Psychotic Attack; Family Members; Acceptance and Commitment Therapy
Keywords: First psychotic attack; family members; Acceptance and Commitment Therapy; group therapy; coping; stigmatization; psychiatric nursing
MeSH Terms: conditions — Stereotyping | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Who Masked: Participant
Masking Description: Experimental: Intervention group ''Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group Intervention: Behavioral: Acceptance and Commitment Therapy No Intervention: Control group Only data collection was carried out. No attempt was made by the researcher during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: ACT (Experimental): ''Acceptance and Commitment Therapy (ACT) Based Intervention Program was applied to the intervention group.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control (No Intervention): Arm Description: Only data collection was carried out. No attempt was made by the researcher during the study.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group in eight sessions online. Each session will last an average of 60-90 minutes. There will be two sessions for one group per week.
  Arms: Experimental: ACT

SUMMARY:
This study aimed to evaluate the effect of ACT administered online to family members on self-stigmatization, coping with stress, and psychological resilience levels after the first psychotic attack (FPA).

DETAILED DESCRIPTION:
This study is a pretest, posttest, follow-up, randomized controlled experimental study. This study will be conducted with family members of individuals diagnosed with FPA who come to the psychiatry outpatient clinic of a training and research hospital. According to the results of G-power analysis, the minimum sample size of the study was calculated as 32 (intervention 16, control 16). Personal Information Form will be applied to the individuals before randomization. The computer-aided https://www.random.org/integers/ program will be used to assign the intervention and control groups without bias. It is planned that the intervention group will consist of 8-12 participants and the program will be implemented as two intervention groups. The Acceptance and Commitment Therapy (ACT) Based Intervention Program will be implemented online in eight sessions. Each session will last 60-90 minutes on average. Two sessions will be held for one group per week. The control group will not receive any intervention from the researcher. The intervention groups will be followed up with a post-test after the program is completed and three months later, while the control group will be followed up with a post-test four weeks and three months later.

In the preparation of the interventions and planning of the sessions based on ACT, the researcher utilized studies in the literature and the basic ACT training she had received. The sessions were prepared based on six components of psychological flexibility found at the basis of ACT.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance to participate in the research,
* Being responsible for the care of an individual who has been diagnosed with schizophrenia and other psychotic disorders according to DSM-5 diagnostic criteria at least six months ago and at most five years ago,
* Living with the patient for at least one year,
* First-degree relatives (mother, father, siblings, adult children and spouse),
* The home environment is suitable for online interviewing (having a computer/smartphone, internet at home, the patient can be alone in the room during the session, etc.),
* Being literate,
* Communication is not a problem.

Exclusion Criteria:

* Refusal to participate in the research,
* Responsible for the care of an individual diagnosed with schizophrenia and other psychotic disorders for less than six months or more than five years according to DSM-V diagnostic criteria,
* Living with the patient for less than one year,
* No first-degree relatives (mother, father, siblings, adult children and spouse),
* The home environment is not suitable for online counseling (having a computer/smartphone, internet at home, the patient can be alone in the room during the session, etc.),
* Illiteracy,
* Communication problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-Stigma Inventory for Families (SSI-F) | 6 month
  The scale was developed to assess the self-stigmatization of family members of individuals diagnosed with schizophrenia. The scores that can be obtained from the scale, which includes 3 factors and 14 items in total, including internalized stereotypes and withdrawal from society, concealment of the disease and perceived worthlessness, vary between 14-70. A high score indicates a high level of self-stigmatization of the family member.

SECONDARY OUTCOMES:
Stress Coping Scale | 6 month
  The scale consists of 23 items and is a 5-point Likert type. It includes 3 sub-dimensions: seeking social support, problem-focused coping and avoidance-focused coping. Items 10, 17 and 20 of the scale are reverse-scored. The total score and subscale scores obtained from the scale provide information about individuals' coping strategies with stress. The scale gives scores ranging from 23 to 115 reflecting the general level of coping strategies used by individuals to cope with stress. High scores obtained from the scale and its subscales indicate an increased tendency to use relevant coping mechanisms.
Brief Resilience Scale | 6 month
  The scale was developed to measure the psychological resilience of individuals. This scale, which consists of 6 items in 5-point Likert type, is a self-report measurement tool. It is scored between "not at all appropriate" (1) and "completely appropriate" (5). Items 2, 4 and 6 of these 6 items are reverse coded. High scores indicate a high level of psychological resilience and low scores indicate a low level of psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Özer, Asst. Prof., Principal Investigator — Bartın Unıversity
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No